CLINICAL TRIAL: NCT06748443
Title: Enhancing Prevention of Injuries in Community (EPIC) Youth and Adult Amateur Football Players - Design of a Type 3 Hybrid Implementation-effectiveness Cluster Randomised Controlled Trial
Brief Title: Enhancing Prevention of Injuries in Community Youth and Adult Amateur Football Players
Acronym: EPIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Collaborators: The Swedish Research Council (Other Government); the Swedish Research Council for Health, Working Life and Welfare (Unknown)
Responsible Party: Principal Investigator, Martin Hägglund, Professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2024-07394-01
Record Dates: First submitted 2024-12-11; First posted 2024-12-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Injury Prevention in Sports; Adherence
Keywords: amateur sports; injury prevention exercise programme; adherence; co-design; support for coaches

STUDY DESIGN:
Intervention Model Description: Type 3 hybrid cluster randomised controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group receiving support for implementation of Knee Control+ (Experimental): Teams in the intervention group will gain access to digital Knee Control+ programme material from the Swedish Football Association website in the pre-season and be introduced to the programme during a digital workshop prior to season start. Additionally, coaches will be offered a smorgasbord of support interventions that they can choose from depending on their specific needs:
  1. physical and digital workshops aiming to increase coach self-efficacy and formalisation of action and coping plans,
  2. site visits to their teams by a study designated fitness coach, aiming to increase coach self-efficacy and player autonomous motivation,
  3. digital programme material with films aiming to increase coach knowledge and inspiration to use Knee Control+,
  4. leaflets about Knee Control+ as inspiration and reminder to use the programme,
  5. social media support as reminder to use the programme.
  Site visits and physical workshops will be led by specifically trained fitness coaches.
  Interventions: Behavioral: Support intervention for the use of Knee Control+; Other: Information about Knee Control+
- Control group with standard introduction of Knee Control+ (Active Comparator): The control group will gain access to the same digital Knee Control+ programme material from the Swedish Football Association website in the pre-season and will be introduced to the programme during a digital workshop prior to study start.
  Interventions: Other: Information about Knee Control+

INTERVENTIONS:
Behavioral: Support intervention for the use of Knee Control+ — Coaches will be offered a smorgasbord of support interventions that they can choose from depending on their specific needs: physical and digital workshops before and during the study, site visits to their team, digital programme material, leaflets and social media posts. Fitness coaches will be responsible for physical workshops to train the football coaches.
  Other Names: Knee Control+; Injury prevention exercise programme
  Arms: Intervention group receiving support for implementation of Knee Control+
Other: Information about Knee Control+ — Coaches receive information about injuries in football and the efficacy of injury prevention exercise programmes at a pre-season digital workshop, and guided to access the Knee Control+ programme from the Swedish Football Association website.

SUMMARY:
This is a type 3 hybrid cluster randomised controlled trial, where implementation of the intervention is the primary outcome and preventive effectiveness is the secondary outcome.

The overall purpose of this study is to evaluate the added value of implementation support on the use and preventive effectiveness of the injury prevention exercise programme Knee Control+ in male and female, youth and adult amateur football teams.

Research questions

1. Does use and injury preventive effect of Knee Control+ differ between teams randomised to an intervention group receiving additional support for Knee Control+ use and teams randomised to a control group with standard access to digital Knee Control+ programme material?
2. Does coach self-efficacy to use Knee Control+, player motivation and player training dosage differ between the intervention and control groups?
3. What are the mediators and moderators that influence use of Knee Control+?
4. How well do the intervention and control groups adhere to Knee Control+ recommended use and is there an association between adherence and preventive efficacy?
5. How are different components of the support material used by the intervention group teams, and how is the implementation support perceived by administrators, coaches and players in the clubs (end-users) and by fitness coaches who educate coaches about the programme (intervention deliverers)?
6. How do coaches perceive their engagement to lead Knee Control+ training with their players and has this changed after having used the implementation support material?

Football teams will be randomised before the 2025 season to an intervention group receiving additional support for the implementation of Knee Control+ or to a control group without this support. All teams will have access to digital programme material via the Swedish Football Association.

Data on implementation of Knee Control+ and injuries (players only) will be collected weekly (coaches) and monthly (players) throughout the season using web-based questionnaires. Behavioural outcomes: for coaches self-efficacy, action and coping planning and perceived support from the club, and for players autonomous motivation, basic psychological needs and basic need support, will also be analysed.

DETAILED DESCRIPTION:
This is a one-season study in the 2025 football season, beginning in the pre-season (March) and ending after the competitive season (November). Football coaches and players are included in the study. A sub-sample of coaches will also be included in a qualitative sub-study after the 2025 season. As part of a process evaluation, club representatives, such as club chairmen, sports directors and youth managers, will also be targeted in the same district, as well as fitness coaches delivering the interventions to the coaches. Coaches will be targeted with most of the interventions, but players and club managers will also benefit from some of the support interventions.

Fitness coaches in a nation-wide organisation (Friskis&Svettis) will be the primary intervention-deliverers and will be educated on the Knee Control+ programme exercises and support interventions to be able to hold workshops at their venues as well as to make site visits in the teams. The research group will be responsible for the education of fitness coaches and will deliver the digital workshops to the coaches and manage the social media account.

Co-design in development of the support material has been employed. During the 2024 season, a working group with representatives for coaches and players (for practical reasons age ≥ 18) was initiated. This working group (two coaches, one former player) provided feedback and new ideas during the development of the support material and the questionnaires for coaches and players.

The workshop concept was tested three times with fitness coaches leading workshops for football coaches during the autumn of 2024 in a district not included in the main study. One site visit was also accomplished and the fitness coaches gave feedback of their experiences to the research group after this.

In the planning and execution of the study, the research group will have regular contact with representatives for football clubs, the district football associations, the Swedish football association and the fitness coach association (Friskis&Svettis) to get their strategic input on the work being done.

Both group constellations have mainly been active during the planning for the study, but some participants may also be invited to give their view on the results and the interpretation of results after the 2025 season. After the 2025 season and potentially before upscaling of the study, the workshop strategies will be followed-up with the fitness coach association and evaluate whether any changes are needed before opening up for national dissemination.

Data will be collected primarily through web-based questionnaires covering implementation outcomes, behavioural outcomes, injury outcomes, adverse events, as well as a process evaluation.

Sample size calculations for the primary outcome were completed using the Shiny CRT online tool for binary outcomes, based on a logistic regression model. Calculations assumed 3 teams per cluster (club); a coefficient of variation equal to 0.9 was applied to account for variation in cluster sizes. An exchangeable correlation structure was assumed, and base case calculations used an intracluster correlation (ICC) of 0.02. Sensitivity analyses considered ICC values between 0.01 and 0.05. The estimated proportion of weeks where teams use the Knee Control+ in the CG is 0.5 (50%), and in the IG 0.8 (80%) based on published data. Considering a design effect (DE) of 1.04, a cluster size of 3 teams will allow for detection of a between-group difference in the primary outcome of at least 0.3 (30%) with 80% power at the 5% level of statistical significance, with total 29 clusters (85 teams). For the same difference in outcome, varying the ICC results between 0.01 and 0.05 rendered sample sizes between 28-30 clusters (83-90 teams). Therefore, the aim is to include minimum 90 teams.

For the main injury outcome, ≥7 days time-loss injuries (secondary outcome), sample size calculations were completed based on a Poisson regression model using the Shiny CRT online tool. Calculations assumed 15 players per team (cluster in the secondary analysis), a coefficient of variation equal to 0.9 was applied to account for variation in cluster sizes. An exchangeable correlation structure was assumed, and base case calculations used an intracluster correlation (ICC) of 0.02. Sensitivity analyses considered ICC values between 0.01 and 0.05. The estimated injury incidence in the CG is 0.2 (20%), and in the IG 0.1 (10%) based on published data. Considering a design effect (DE) of 1.28, a cluster size of 15 players will allow detection of a between-group relative difference in the secondary outcome of at least 0.5 (50% injury reduction) with 80% power at the 5% level of statistical significance, with total 41 teams (607 players). For the same difference in outcome, varying the ICC results between 0.01 and 0.05 rendered sample sizes between 37-54 teams (541-806 players). This equals to total 14 clusters (range 12-18 clusters) at a club level.

Data on any football related injury will be collected regardless of need of care or absence from football training or matches ("all physical complaints" injury definition).

The primary outcome, use of Knee Control+, will be analysed at team-level as the proportion of weeks with sufficient use of the programme and compared between intervention group and control group using logistic regression. The limit for sufficient training frequency is set at Knee Control+ training at least 2 times per week. Since a gradual start of injury prevention training is preferred for beginners, for players 10-12 years use of ≥3 of 6 main exercises is deemed sufficient, whereas for players >12 years, use of ≥4 of 6 main exercises is deemed sufficient to be defined as use of Knee Control+. Other measures of implementation will also be compared between groups and predominantly with parametric statistics.

Injury incidence rate (injuries per 1000 athlete exposures) and monthly prevalence rate (number of injured athletes/total number of athletes each month) will be presented with 95% confidence intervals, and incidence rate ratio and prevalence rate ratio will be calculated and compared between groups (according to intention-to-treat) using Generalized Linear Models with Poisson distribution, log link and the natural logarithm of total athlete exposures or total eligible weeks as offset denominator variables.

Qualitative interviews will be analysed using qualitative content analysis and an inductive approach.

ELIGIBILITY:
Inclusion Criteria:

* Male and female, youth and adult amateur football teams
* Teams participating in series for players 10 years or older
* Teams with scheduled training at least twice per week during the season
* All eligible players in the team are invited to participate, regardless of whether they have an injury or not at study start

Exclusion Criteria:

* Players with long-term injuries not planning to take part in match play in the 2025 season

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Use of Knee Control+ | One season, 7 months, from start of the competitive season (April 2025) to the end of the competitive season (October 2025)
  Proportion of weeks in the season with Knee Control+ training being performed at least 2 times in that week with sufficient completion of Knee Control+ components: for players 10-12 years, use of at least 3 of 6 main exercises OR for players >12 years, use of at least 4 of 6 main exercises, as reported by coaches in a web-based questionnaire on a weekly basis.

SECONDARY OUTCOMES:
Adherence to Knee Control+, cumulative utilisation | Reported weekly during the 7 months competitive season (April-October 2025)
  Proportion of training sessions where Knee Control+ was used, registered by coaches
Adherence to Knee Control+, utilisation frequency | Reported weekly (coaches) or monthly (players) during the 7 months competitive season (April-October 2025), as well as at follow-up 1 week after the season (November 2025)
  Use of Knee Control+ n times/week
Adherence to Knee Control+, duration fidelity | Reported at follow-up 1 week after the season (November 2025)
  Minutes spent on Knee Control+ each session, reported by coaches
Adherence to Knee Control+, utilisation fidelity | Reported at follow-up 1 week after the season (November 2025)
  Assessed using questions about how Knee Control+ was used at training. Reported by coaches and players.
Behavioural outcomes, self-efficacy | Reported by coaches at baseline (March 2025), monthly during the 7 months competitive season (April-October 2025) and follow-up 1 week after the season (November 2025)
  Change in perceived self-efficacy from baseline to follow-up. Three questions about action self-efficacy based on the Health Action Process Approach (numerical rating scale 0-10, where 0 is the least and 10 the most favorable option. Exercise self-efficacy with the Exercise Self-Efficacy Scale (9 questions, numerical rating scale 0-10, where 0 is equal to "not confident at all" and 10 is equal to "completely confident", i.e. 0 is the least and 10 is the most favourable option).
Behavioural outcomes, presence of action plans | Reported at baseline (March 2025) and follow-up 1 week after the season (November 2025), as well as mid-season (August 2025).
  One question based on the Health Action Process Approach, reported by coaches, rated on a numerical rating scale 0-10, where 0 is the least and 10 the most favourable option. Comparison of presence of action plans between groups.
Behavioural outcomes, presence of coping plans | Reported at mid-season (August 2025) and at follow-up 1 week after the season (November 2025)
  One question based on the Health Action Process Approach, reported by coaches and rated on a numerical rating scale 0-10, where 0 is the least and 10 the most favourable option. Comparison of presence of coping plans between groups.
Behavioural outcomes, perception of club support | Reported at follow-up 1 week after the season (November 2025)
  Reported by coaches using the General Training Climate Scale (6 questions, Likert 1-5, where 1 is the least and 5 the most favourable option). Compared between groups.
Behavioural outcomes, autonomous and controlled motivation | Reported at baseline (March 2025) and follow-up 1 week after the season (November 2025)
  Change in autonomous versus controlled motivation. Reported by players with the Treatment Self-Regulation Questionnaire (4 questions focusing on autonomous motivation on a Likert 1-7, where 1 represent less and 7 more autonomous motivation, 4 questions focusing on controlled motivation on a Likert 1-7, where 1 represent less and 7 more controlled motivation).
Behavioural outcomes, basic psychological needs | Reported at mid-season (August 2025) and follow-up 1 week after the season (November 2025)
  Reported by players using single-items scales (3 questions, Likert scale 1-7, where 1 is the least and 7 the most favourable option). Compared between groups.
Behavioural outcomes, basic need support | Reported at follow-up 1 week after the season (November 2025)
  Reported by players using the Coaching Behavior Scale for Sport and specifically the construct covering technical skills (7 questions, Likert scale 1-7, where 1 is the least and 7 the most favourable option). Compared between groups.
Injury outcomes, incidence of new injuries | Reported monthly during the 7 months competitive season (intervention period, April-October 2025).
  Reported by players using the Oslo Sports Trauma Research Center Overuse Injury Questionnaire (OSTRC-O2, 4 questions) and additional questions to specify the injury. Injury incidence is presented separately for three severity categories:
  1. ≥7 days time-loss injuries (primary injury outcome variable is 7 day time-loss injury to the lower extremity),
  2. time-loss injuries (secondary injury outcome variable),
  3. all injuries (secondary injury outcome variable)
Injury outcomes, monthly prevalence of injuries | Reported monthly during the 7 months competitive season (intervention period, April-October 2025).
  Reported by players using the Oslo Sports Trauma Research Center Overuse Injury Questionnaire (OSTRC-O2, 4 questions) and additional questions to specify the injury. Injury prevalence is presented separately for three severity categories:
  1. ≥7 days time-loss injuries,
  2. substantial injuries (moderate or severe modifications in football participation and/or moderate or severe effects on football performance, or inability to participate in football,
  3. all injuries
Adverse events | Reported at follow-up 1 week after the season (November 2025)
  Coaches and players will report on any adverse events related to the training intervention Knee Control+. 3 bespoke questions about occurrence, frequency and type of adverse event.

OTHER OUTCOMES:
Process evaluation, number of teams that participate in physical workshops | Reported at follow-up 1 week after the season (November 2025)
  N teams (intervention group) that have taken part in workshops.
Process evaluation, number of teams that participate in site visits | Reported at follow-up 1 week after the season (November 2025)
  N teams that have had a fitness coach visiting their team
Process evaluation, number of teams that participate in booster workshops | Reported at follow-up 1 week after the season (November 2025)
  N teams (intervention group) that have taken part during workshops
Process evaluation, number of teams that participate in digital workshops | Reported at follow-up 1 week after the season (November 2025)
  N teams (intervention group) that have taken part during digital workshops
Process evaluation, number of teams that use printed programme material | Reported at follow-up 1 week after the season (November 2025)
  N teams (intervention group) that have used the printed programme material
Process evaluation, number of teams that use digital programme material | Reported at follow-up 1 week after the season (November 2025)
  N teams (intervention group) that have used digital programme material
Process evaluation, number of teams that use social media account | Reported at follow-up 1 week after the season (November 2025)
  N teams (intervention group) that have followed the study specific social media account
Process evaluation, number of teams that use Knee Control+ material via the Swedish Football Association | Reported at follow-up 1 week after the season (November 2025)
  N teams (control and intervention group) that have used the programme material
Process evaluation, perceptions of the support intervention (quantitative) | Reported at follow-up 1 week after the season (November 2025), and immediately after taking part in workshops or site visits during the 7 months competitive season (April-October 2025)
  Bespoke questionnaire, with questions on a numerical rating scale 0-10, where 0 is the least and 10 the most favourable option, distributed to coaches (and in relevant cases players) after taking part in workshops or site visits
Process evaluation, perceptions of the support intervention (qualitative) | Reported in qualitative sub-study after the season (November 2025-March 2026)
  Assessed during qualitative interviews with coaches
Process evaluation, web statistics | Assessed throughout the study (from pre-season March 2025, competitive season April-October 2025, until follow-up 1 week after the season in November 2025)
  Access and use of different modules in digital intervention material. Number of unique visits to the web page.
Process evaluation, club prevention policies and practices | Reported at follow-up 1 week after the season (November 2025)
  Reported by club representatives using a bespoke questionnaire (12 questions, numerical rating scale 0-10, where 0 is the least and 10 the most favourable option, and open-ended questions).
Process evaluation, perceptions about the education of coaches | Reported at follow-up 1 week after the season (November 2025)
  Reported by fitness coaches in a bespoke questionnaire (12 questions, numerical rating scale 0-10, where 0 is the least and 10 the most favourable option, and open-ended questions).

CONTACTS AND LOCATIONS:
Overall Officials: Martin Hägglund, Professor, Principal Investigator — Linköping university, Department of Health, Medicine and Caring Sciences, Unit of Physiotherapy
Locations (1):
- Linköping university, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data that underlie results in publications may be available upon reasonable request to the principal investigator
Supporting Information: Study Protocol
Time Frame: 1 year after publication
Access Criteria: De-identified individual participant data that underlie results in publications may be available upon reasonable request to the principal investigator

REFERENCES:
- [Derived] Lindblom H, Sonesson S, Walden M, Akerlund I, Ivarsson A, Hagglund M. Enhancing Prevention of Injuries in Community youth and adult amateur football teams (EPIC) via implementation support for an exercise-based intervention: study protocol for a type 3 hybrid implementation-effectiveness cluster-randomised controlled trial. BMJ Open. 2025 Aug 26;15(8):e102008. doi: 10.1136/bmjopen-2025-102008. PMID 40858379